CLINICAL TRIAL: NCT04765592
Title: Guo's Aortic Arch Reconstruction :The Prospective ,Multiple Center Study About the Safety and Efficacy of WeFlow-Arch Modeler Embedded Branch Stent Graft System (GIANT Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEIQIANG202001
Record Dates: First submitted 2021-02-04; First posted 2021-02-21 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Aortic Arch Aneurysm
MeSH Terms: conditions — Aneurysm, Aortic Arch

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WeFlow-Arch Modeler Embedded Branch Stent Graft System (Experimental): Participants will be treated with WeFlow-Arch Modeler Embedded Branch Stent Graft System
  Interventions: Device: WeFlow-Arch Modeler Embedded Branch Stent Graft System

INTERVENTIONS:
Device: WeFlow-Arch Modeler Embedded Branch Stent Graft System — The modular embedded aortic arch stent graft system consists of the embedded ascending aorta stent graft system, the arch aorta stent graft system and the branch stent system.

SUMMARY:
A prospective ,Multiple Center Study About the Safety and Efficacy of WeFlow-Arch Modeler Embedded Branch Stent Graft System manufactured by EndoNom Medtech (Hangzhou) Co., Ltd. for true/false aortic arch aneurysms and ulcers involving aortic arch . (GIANT Study)

DETAILED DESCRIPTION:
This study is a prospective ,multiple center study about the safety and efficacy of WeFlow-Arch Modeler Embedded Branch Stent Graft System, it is expected to complete the implantation of 80 patients in 23 centers within 12 months, and interim follow-up was conducted before discharge, 30 days after surgery, 6 months after surgery and 12 months after surgery, long-term follow-up will be performed at 24 months postoperatively, 36 months postoperatively, 48 months postoperatively and 60 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years old;
2. Diagnosed with aortic arch lesions requiring intervention, including true aortic arch aneurysms, pseudo-aortic arch aneurysms, and ulcers involving the aortic arch;
3. Showing a suitable vascular condition, including:

   * Ascending aorta length greater than 50 mm (from the aortic sinusoid junction to the proximal cardiac margin of the innominate artery).
   * Ascending aorta diameter ≥ 24 mm and ≤ 48 mm;
   * Proximal anchoring zone length ≥ 30 mm;
   * Innominate artery diameter ≤ 24 mm and ≥ 7 mm, length ≥ 20 mm；
   * Left common carotid artery or left subclavian artery diameter ≤ 24 mm and ≥ 7 mm, length ≥ 20 mm；
   * Suitable arterial access for endovascular interventional treatment;
4. Able to understand the purpose of the trial, participate in the trial voluntarily with informed consent form signed by the patient him/herself or his or her legal representative, and willing to complete follow-up visits as required under the protocol.
5. Evaluated by at least two vascular surgeons or cardiac surgeons as high surgical risk patients or deemed to have significant surgical contraindications.

Exclusion Criteria:

1. Experienced systemic infection during past three months;
2. Neck surgery was performed within 3 months;
3. Previous endovascular interventional treatment involving the aortic arch was performed;
4. Infectious aortic disease、Takayasu arteritis，Marfan syndrome (or other connective tissue diseases );
5. Severe stenosis, calcification, thrombosis, or tortuosity of the carotid or subclavian artery;
6. Heart transplant;
7. Suffered MI or stroke during past three months;
8. Class IV heart function (NYHA classification);
9. Active peptic ulcers or upper gastrointestinal bleeding occurring within the previous three months;
10. Hematological abnormality, defined as follows: Leukopenia (WBC < 3 × 109/L), acute anemia (Hb < 90 g/L); thrombocytopenia (PLT count < 50 × 109/L), history of bleeding or coagulopathy;
11. Renal insufficiency， creatinine > 265 umol/L (or 3.0mg/dL) and/or end-stage renal disease requiring renal dialysis, as determined by an investigator after a thorough analysis;
12. Pregnant or breastfeeding;
13. Allergies to contrast agents;
14. Life expectancy of less than 12 months;
15. Participating in another drug or device research;
16. Any other disease or abnormality that the investigators believe may hinder endovascular interventional treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2025-02-05 (Estimated); Study Completion 2029-02-05 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality and major stroke within 12 months after surgery | 12 months after surgery
  All-cause mortality includes cardiac mortality, non-cardiac mortality, and mortality from unknown causes. Severe stroke is defined as a modified Rankin score (mRS) ≥ 2 at 90 days following stroke onset.

SECONDARY OUTCOMES:
Rate of immediate technical success following surgery | immediately after the surgery
  Immediate technical success is defined as successful delivery of the aortic and branching stent graft conveyors to their predetermined positions, accurate positioning and successful deployment of the stent, safe removal of the delivery device outside the body, and the absence of Type I and III endoleaks per imaging studies conducted at the end of the procedure with all branching stents patency.
Rate of aortic aneurysm progression under control | 12 months after operation
  Aortic aneurysm progression under control is defined as maximum increase in the diameter of the aortic aneurysm was ≤ 5 mm when compared with preoperative aortic aneurysm as of a 12-month postoperative CTA review
Incidence of Type I or Type III endoleak | immediately after the surgery, 1 month, 6 months, 12 months after the surgery
  Incidence of Type I or Type III endoleak before discharge, 1 month, 6 months, 12 months after operation. Intraoperative endoleaks subject to adjuvant treatment are not recorded. Endoleaks occurring after the completion of the procedure followed by one or more endoleaks occurring in the same subject at different follow-up stages that were not treated are counted as a single instance.
Incidence of aortic arch stent graft displacement | 1 month, 6 months, 12 months after operation
  CTA examination will be performed at 1 month, 6 months, and 12 months post operation to determine if the stent has migrated, and evaluations will be recorded for both the main and branch stents. Displacement is defined as a nodal aortic or branching stent graft displacement of more than 10 mm from pre-discharge levels.
Postoperative branch vessel patency rate | 1 month, 6 months, 12 months after operation
  CTA examinations will be performed at 1 month, 6 months, and 12 months post operation to evaluate branch vessel reconstruction and assess for occlusion, stenosis, or in-stent thrombosis.
Incidence of surgically induced de novo aortic dissection converted to open-heart surgery or secondary intervention | 30 days, 6 months, and 12 months after operation
  Incidence of surgically induced de novo aortic dissection converted to open-heart surgery or secondary intervention 30 days, 6 months, and 12 months after operation.Whether or not the patient experienced surgically induced de novo aortic dissection converted to open-heart surgery or secondary intervention will be determined.
Rate of major adverse events | 30 days post operation
  Refers to all-cause mortality, myocardial infarction, ischemic stroke, or respiratory failure occurring within 30 days after surgery. More specifically, myocardial infarction refers to a drastic reduction or complete interruption of the coronary blood supply due to coronary artery disease, resulting in severe and prolonged acute ischemia of the corresponding myocardium, leading to necrosis of cardiomyocytes. Ischemic stroke refers to the result of necrosis of brain tissue caused by narrowing or occlusion of the arteries supplying blood to the brain or insufficient blood supply to the brain. Respiratory failure is defined as a state resulting in significantly prolonged intubation, tracheotomy, deterioration of lung function, or other fatal outcomes.
Rate of aortic aneurysm-related mortality | 12 months post operation
  Refers to mortality caused by a ruptured aortic aneurysm or endovascular interventional treatment.
Incidence of severe adverse events | 30 days, 6 months, and 12 months after operation
  Refers to an event that occurs during the clinical trial that results in mortality or serious deterioration in patient health, including a fatal illness or injury, a permanent defect in body structure or body function, or an event that requires medical or surgical intervention to avoid one or more permanent defects in body structure or body function.
Incidence of device-related adverse events | 30 days, 6 months, and 12 months after operation
  Device-related adverse events refer to an adverse medical event related to the use of a device that occurs during the clinical trial. However, a distinction should be made with respect to normal postoperative stress response, such as fever and chest and back discomfort, which, in the judgment of the investigator, need not be recorded as an adverse event. Recording of device-related adverse events will be applicable for conditions that are deemed by the investigator to be definitely related, possibly related, or of indeterminate relationship, to the test device.

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Chinese PLA General Hospital, Beijing
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University People's Hospital, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital ,Sun Yat-sen University, Guangzhou
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - Shandong Provincial Hospital, Jinan
  - The First People's Hospital of Yunnan Province, Kunming
  - Nanjing Drum Tower Hospital, Nanjing
  - Nanjing First Hospital, Nanjing
  - The Affiliated Hospital Of Qingdao University, Qingdao
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - The Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai
  - The First Affiliated Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital Of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of PLA Air Force Military Medical University, Xi'an
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared for scientific purposes after the completion of the clinical trial. However, patients' electronic records and any CTA files are outside the scope of our data sharing policy. Researchers wanting to request data can submit a detailed application to the investigators. Data will be released depending on the scientific quality of the submitted request.
Supporting Information: Study Protocol, ICF
Time Frame: It is expected that data will be obtained after study completion for at least one year.

REFERENCES:
- [Derived] Liu F, Zhang H, Rong D, Ge Y, Jia X, Xiong J, Ma X, Wang L, Fan T, Guo W. Protocol for Guo's aortIc Arch recoNstrucTion: a prospective, multicentre and single-arm study to evaluate the safety and efficacy of the WeFlow-Arch modular inner branch stent-graft system for aortic arch lesions (GIANT study). BMJ Open. 2022 Oct 10;12(10):e063245. doi: 10.1136/bmjopen-2022-063245. PMID 36216431